CLINICAL TRIAL: NCT06439862
Title: Quality of Life in School Aged-children With Posterior Urethral Valves
Brief Title: Study of the Quality of Life in School Aged-children With Posterior Urethral Valves
Acronym: QUALIVUP
Status: Recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL24_0181
Record Dates: First submitted 2024-05-28; First posted 2024-06-03 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Quality of Life; Posterior Urethral Valve; Renal Insufficiency; Chronic Renal Disease; End Stage Renal Disease; Bladder Dysfunction; Urinary Incontinence
Keywords: Quality of life; Posterior Urethral Valves; Children; Adolescents; Family
MeSH Terms: conditions — Renal Insufficiency; Renal Insufficiency, Chronic; Kidney Failure, Chronic; Urinary Incontinence

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Children with PUV — Male children aged 6 to 17 years old treated for PUV in their first year of life between 2006 and 2018 in Lyon, and managed in the Femme-Mère-Enfant Hospital in Lyon

SUMMARY:
Posterior urethral valves (PUV) are the most common congenital obstructive lesion of the urethra, affecting from 1 per 3000 to 1 per 8000 live births. Valve ablation usually resolves the obstruction in PUV but patients still may suffer of deterioration in renal and urinary functions.

Renal insufficiency is the most feared long-term complication. Up to 50 % of the patients will develop chronic kidney disease (CKD), and up to 20 % will develop end-stage renal disease (ESRD) and ultimately will require kidney transplantation. PUV is the first urological cause of ESRD. Progression towards CKD depends on febrile urinary tract infections (UTIs), severity of a vesicoureteral reflux and bladder dysfunction.

Bladder dysfunction is due to an overactive and small poorly compliant bladder during infancy. Detrusor overactivity usually decreases in childhood and bladder capacity increases. The most common symptom of this bladder dysfunction is urinary incontinence. 60 % of children are continent at the age of 5 years old and 90 % at 10 years old. In case of persistent bladder dysfunction, medical treatment (anticholinergics, alpha-blockers) may be introduced, or even intermittent catheterizations.

Current scientific literature has very few studies on quality of life (QoL) in patients with PUV, mostly in adult patients and very small cohorts. Men treated for PUV in childhood had a good quality of life compared to the normative population, except for sleeping, eating and sexual activity. It seemed that the more severe the urological and nephrological functions were, the lower the QoL was. Children were only asked about intermittent urinary catheterization, and family point of view has never been collected. However, QoL and long-term evolution represent the first concerns of parents-to-be in prenatal counseling, or after diagnosis in an infant with PUV.

Hence, the aim of the study is to investigate the quality of life in school-aged children who had been treated for PUV in their first year of life, as measured by the Pediatric Quality of Life Inventory Version 4.0 (PedsQL 4.0).

ELIGIBILITY:
Inclusion Criteria:

* Male patients and their parents/relatives
* Aged 6 to 17 years old
* Treated for PUV in their first year of life between 2006 and 2018
* Managed in the Femme-Mère-Enfant Hospital in Lyon

Exclusion Criteria:

* Children with pre-existing severe cognitive and physical disability (physician's rating) from other condition
* Children enable to complete QoL questionnaire due to mental or communication impairment

Ages: 6 Years to 17 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with PUV will be selected inside the database of the pediatric surgery department of the Femme-Mère-Enfant Hospital in Lyon
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-08-20 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Score of the PedsQL 4.0 (Pediatric Quality of Life Inventory Version 4.0) Generic Core Scales | At inclusion
  The PedsQL 4.0 measures health-related quality of life in healthy children and those with acute and chronic health conditions. It consists of parallel child self-report and parent proxy-report formats, with 23 items and 5 response selections that range from "never" to "almost always". Parent proxy-report assesses parent's perceptions of their child's HRQOL. The items for each of the forms are essentially identical, differing in developmentally appropriate language, or first or third person tense.
  Items are reverse-scored and linearly trans-formed to a 0 to 100 scale (0 = 100, 1 = 75, 2 = 50, 3 = 25, 4 = 0), so that higher scores indicate better HRQOL. Scale Scores are computed as the sum of the items divided by the number of items answered (this accounts for missing data). If more than 50% of the items in the scale are missing, the Scale Score is not computed.

CONTACTS AND LOCATIONS:
Overall Officials: BIDAULT Valeska, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Femme-Mère-Enfant Hospital, Bron, Bron, France

IPD SHARING:
Plan to Share IPD: No